CLINICAL TRIAL: NCT01531465
Title: Pulmonary Function Testing in Infants With Respiratory Insufficiency While Receiving High Flow Nasal Cannula (HFNC) Versus Nasal Continuous Positive Airway Pressure (nCPAP)
Brief Title: High Flow Nasal Cannula Versus Nasal Continuous Positive Airway Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christiana Care Health Services (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 31073
Record Dates: First submitted 2011-05-25; First posted 2012-02-13 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Respiratory Insufficiency
Keywords: Respiratory insufficiency; Infants; High Flow Nasal Cannula (HFNC); Nasal Continuous Positive Airway Pressure (NCPAP)
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Respiratory Physiological Phenomena

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HFNC to NCPAP (Other): Infants who are currently on HFNC.
  Interventions: Other: Pulmonary function testing and esophageal pressure
- NCPAP to HFNC (Other): Infants who are currently on NCPAP.
  Interventions: Other: Pulmonary Function Testing & esophageal pressure monitoring

INTERVENTIONS:
Other: Pulmonary Function Testing & esophageal pressure monitoring — Infants who are currently on NCPAP will have pulmonary function testing (PFTs)and esophageal pressure performed while on 2 different settings of NCPAP. These infants will then be transitioned HFNC and will undergo PFTs and esophageal pressure while on different HFNC settings. The infant will then be returned to NCPAP at the same settings they were on prior to any study interventions.
  Other Names: Pulmonary Function Testing; Esophageal pressure
  Arms: NCPAP to HFNC
Other: Pulmonary function testing and esophageal pressure — Infants who are currently on HFNC will have pulmonary function testing (PFTs) and esophageal pressure performed while on 2 different settings of HFNC. These infants will then be transitioned NCPAP and will undergo PFTs and esophageal pressure while on 2 different NCPAP settings. The infant will then be returned to HFNC at the same settings they were on prior to any study interventions.
  Other Names: Pulmonary Function Testing; Esophageal pressure
  Arms: HFNC to NCPAP

SUMMARY:
The purpose of this study is to compare two common methods of providing respiratory support: nasal continuous airway pressure and high flow nasal cannula to see what effect it has on babies breathing. The investigators also will compare the effects of slightly changing the level of support these two different types of therapy on how easily your baby is breathing. Changes in the level of support and between these two respiratory support modalities are frequently done and are part of the routine care in the neonatal intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* Infants who are between 28 and 40 weeks of corrected gestational age at the time of study entry
* Currently on high flow nasal cannula receiving 3 to 5 lpm or on nasal continuous positive airway pressure at 5 to 6 cmH2P with and FiO2 requirement </= 40% by the clinical care team for clinical care purposes.
* On current mode of support for >/= 12 hours and have been extubated from a mechanical ventilator for >/= 48 hours.

Exclusion Criteria:

* Infants with skeletal or neuromuscular disorders that affect the accuracy of RIP PFT measurements.

Ages: 2 Days to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2011-06; Primary Completion 2012-10 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
lung compliance | 2 hours
  Is there a difference in pulmonary function tests in infants with respiratory insufficiency being treated with high flow nasal cannula (HFNC) or nasal continuous positive airway pressure (NCPAP)?

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz de Jongh, MD, Principal Investigator — Christiana Care Health Systems; Robert Locke, DO, Study Director — Christiana Care Health Services
Locations (1):
- Christiana Care Health System - Christiana Hospital, Newark, Delaware, United States